CLINICAL TRIAL: NCT01125306
Title: Efficiency of XAL-EASE Device in Glaucoma and/or Ocular Hypertension (OHT) Patients, Treated With Xalatan or Xalacom
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLAUCOMA/XAL EASE 1
Record Dates: First submitted 2010-05-16; First posted 2010-05-18 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Glaucoma; Hypertension
Keywords: Drug consumption; The Xal-Ease device; Patient's compliance; Using a novel Pfizer-Pharmacia device to facilitate the Xalatan/Xalacom instillation and to avoid loss of eye drops
MeSH Terms: conditions — Glaucoma; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Xal-Ease — Xal-Ease device used to facilitate application of Xalatan/Xalacom eye drops.
  Other Names: Xal-Ease as a Pfizer-Pharmacia device.

SUMMARY:
Xal-Ease is a novel Pfizer-Pharmacia device aimed to significantly facilitate the Xalatan/Xalacom instillation and to avoid loss of Xalatan/Xalacom eye drops due to incorrect instillation.

Patients on Xalatan/Xalacom who have consumed more than one bottle per month within a year according to consumption data drawn from the Clalit Health Services database, will use the Xal-Ease device for a year. The device is expected to reduce consumption of bottles and result in saving money for both patients and medical care providers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma or hypertension treated with Xalatan/Xalacom who have consumed more than one bottle per month within a year prior to initiation of the study.

Exclusion Criteria:

* Patients younger than 18 years,
* Patients with severe manual disabilities,
* Patients with impaired cognition and mentality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Consumption of Xalatan/Xalacom bottles per year per patient. | 12 months.

SECONDARY OUTCOMES:
Evaluating cost of Xalatan/Xalacom eye drops use per year with Xal-Ease | 12 months
Characterizing the optimal conditions for proper usage of the Xal-Ease device | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology department, Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Semes L, Shaikh AS. Evaluation of the Xal-Ease latanoprost delivery system. Optometry. 2007 Jan;78(1):30-3. doi: 10.1016/j.optm.2006.06.016. PMID 17208672
- [Result] Nordmann JP, Baudouin C, Bron A, Denis P, Rouland JF, Sellem E, Renard JP. Xal-Ease: impact of an ocular hypotensive delivery device on ease of eyedrop administration, patient compliance, and satisfaction. Eur J Ophthalmol. 2009 Nov-Dec;19(6):949-56. doi: 10.1177/112067210901900609. PMID 19882583
- See also: Related Info — http://www.xalatan.com/tools/xal-ease.aspx